CLINICAL TRIAL: NCT07049835
Title: A Double-Blind Randomized Controlled Trial of Ilioinguinal Nerve Block With Local Anesthetic vs. Placebo in Inguinal Hernia Repair Under Spinal Anesthesia
Brief Title: Ilioinguinal Nerve Block With Local Anesthetic vs. Placebo in Inguinal Hernia Repair Under Spinal Anesthesia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Mohamad-Ali Barada, Anesthesia Attending, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MGH-06-25017
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Inguinal Hernias
Keywords: Bupivacaine Hydrochloride; Spinal Anesthesia; Nerve Blocks; Iliohypogastric Nerve Neuralgia; Ilioinguinal Neuralgia; Adults; Lidocaine Hydrochloride; Normal Saline; Sulfentanyl
MeSH Terms: conditions — Hernia, Inguinal; Neuralgia

STUDY DESIGN:
Intervention Model Description: This study will be a randomized prospective , double-blind, controlled trial conducted in a tertiary care surgical unit.
  A total of 100 patients (50 in each group) undergoing lower Inguinal hernia surgery will be enrolled based on power analysis.
  Anesthetic Technique
  * Group A: Spinal anesthesia will be administered using a standard technique with a 25G spinal needle, targeting the appropriate vertebral level.
  * Group B: In addition to spinal anesthesia, an ultrasound-guided ilioinguinal nerve block will be performed post to the surgical incision.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Mixture Block (Active Comparator): 15cc 0.25% of Bupivacaine + Dexamethasone 8 mg 2cc
  Interventions: Drug: Ilioinguinal/iliohypogastric Nerve Block
- Intrathecal Placebo (Placebo Comparator): 17 cc of Ns/s
  Interventions: Other: Ilioinguinal/iliohypogastric with Placebo Block

INTERVENTIONS:
Drug: Ilioinguinal/iliohypogastric Nerve Block — 15cc 0.25% of Bupivacaine + Dexamethasone 8 mg 2cc
  Arms: Intrathecal Mixture Block
Other: Ilioinguinal/iliohypogastric with Placebo Block — 17 cc of Placebo
  Arms: Intrathecal Placebo

SUMMARY:
Postoperative pain management remains a critical area of concern in surgical practices, especially in procedures involving the lower abdomen and pelvis. Inguinal Hernia is considered among few surgeries that may lead to chronic pain. Spinal anesthesia is a commonly utilized modality because of its efficacy in pain control and rapid recovery. However, the addition of peripheral nerve blocks, such as the ilioinguinal nerve block, may provide enhanced pain relief and reduce opioid consumption postoperatively. This study aims to evaluate the effectiveness of spinal anesthesia alone compared to spinal anesthesia supplemented with ultrasound-guided ilioinguinal and iliohypo-gastric nerve block in managing postoperative pain.

DETAILED DESCRIPTION:
Objectives

1. Primary Objective: To compare the postoperative pain scores (using a standardized numerical rating scale) between patients receiving spinal anesthesia alone and those receiving spinal anesthesia with ultrasound-guided ilioinguinal nerve block.
2. Secondary Objectives:

   * To assess the total opioid consumption in the first 24 hours post-surgery.
   * To evaluate the time to first analgesic request postoperatively.
   * Patient Satisfaction score post-op >> at rest , coughing , ambulation ( LEKENT SCORE ) .

Hypotheses

* Hypothesis 1: Patients receiving spinal anesthesia with an ilioinguinal nerve block will experience significantly lower postoperative pain scores compared to those receiving spinal anesthesia alone.
* Hypothesis 2: Patients receiving spinal anesthesia with an ilioinguinal nerve block will require less opioid medication in the first 24 hours post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* ASA physical status I-III
* Scheduled for elective lower abdominal surgery (e.g., inguinal hernia repair, cesarean section)

Exclusion Criteria:

* Allergy to local anesthetics
* Coagulation disorders
* Infection at the injection site
* Patients with neurological conditions affecting lower limbs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain management | 24 hours
  Pain scores will be assessed using an 11-point numerical rating scale (0-10) at 1, 6, 12, and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmazlar A, Bilgel H, Donmez C, Guney A, Yilmazlar T, Tokat O. Comparison of ilioinguinal-iliohypogastric nerve block versus spinal anesthesia for inguinal herniorrhaphy. South Med J. 2006 Jan;99(1):48-51. doi: 10.1097/01.smj.0000197298.48311.80. PMID 16466122
- [Background] Zhou Y, Chen M, Zhang Y, Zhou H, Yu X, Chen G. Ilioinguinal/iliohypogastric nerve block versus transversus abdominis plane block for pain management following inguinal hernia repair surgery: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2019 Oct;98(42):e17545. doi: 10.1097/MD.0000000000017545. PMID 31626118